CLINICAL TRIAL: NCT00469287
Title: Exploration of Early Diagnosis of Diabetes Mellitus Type 2 Based on Traditional Chinese Medicine by MERID Diagnostics, Biophoton Measurements, Heart Rate Variability and Systems Biology
Brief Title: Early Diagnosis of Diabetes Mellitus Type 2 (DM2)
Acronym: 7348
Status: Completed | Type: Observational
Sponsor: TNO (Other)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government)
Responsible Party: Dr. W.J. Pasman, TNO Quality of Life
Other Study IDs: P7348
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2008-04-07 (Estimated); Status verified 2008-04

CONDITIONS: Impaired Blood Glucose Level; Overweight; Obesity
Keywords: diabetes mellitus; blood sugar; overweight; obesity; Traditional Chinese medicine
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Rationale: The global prevalence of diabetes, along with its devastating effects on life expectancy and quality of life, continues to increase. Worldwide, the total number of people with diabetes is projected to rise from about 171 million in 2000 to 336 million in the year 2030. Type 2 diabetes accounts for about 85 percent to 95 percent of all diagnosed cases of diabetes and is associated with a number of serious long-term complications, which are a major cause of morbidity, hospitalization and mortality in diabetic patients. More evidence is becoming available that both lifestyle and clinical intervention in the pre-diabetic condition are effective in slowing down progression of pre-diabetes to overt diabetes.

Over many centuries, several forms of traditional medicine have developed which are often based on fundamental principles that differ from those of "Western" medicine. One of the most prominent characteristics of Traditional Chinese Medicine (TCM), is a more holistic approach to the functioning and disfunctioning of living organisms. Every healthy organism is in a Yin Yang balance and is considered to be a complex interplay between body and mind. Western medicine relies on detailed classification of diseases, empirical investigations and treatments targeting those disorders. However, "Western medicine" is showing an increased interest in traditional forms of medicine.

Objectives: The primary objective of the present study is to determine consistency in classification of DM type 2 in three categories as defined by Traditional Chinese Medicine (TCM) in pre-diabetic subjects.

Secondary objectives are to find relationships between diagnosis according to TCM and risk profile according to Western approach (fasting glucose and HbA1c in plasma, age, BMI, waist circumference). Another objective is to find relationships between classification of risk for DM type 2 according to TCM and objective parameters.

DETAILED DESCRIPTION:
Rationale: The global prevalence of diabetes, along with its devastating effects on life expectancy and quality of life, continues to increase. Worldwide, the total number of people with diabetes is projected to rise from about 171 million in 2000 to 336 million in the year 2030. Type 2 diabetes accounts for about 85 percent to 95 percent of all diagnosed cases of diabetes and is associated with a number of serious long-term complications, which are a major cause of morbidity, hospitalization and mortality in diabetic patients. More evidence is becoming available that both lifestyle and clinical intervention in the pre-diabetic condition are effective in slowing down progression of pre-diabetes to overt diabetes.

Over many centuries, several forms of traditional medicine have developed which are often based on fundamental principles that differ from those of "Western" medicine. One of the most prominent characteristics of Traditional Chinese Medicine (TCM), is a more holistic approach to the functioning and disfunctioning of living organisms. Every healthy organism is in a Yin Yang balance and is considered to be a complex interplay between body and mind. Western medicine relies on detailed classification of diseases, empirical investigations and treatments targeting those disorders. However, "Western medicine" is showing an increased interest in traditional forms of medicine.

The progress in research, especially metabolomics, as the ultimate phenotyping, has been shown to enable the efficacy study of complex mixtures such as Traditional Chinese Medicine (TCM) in complex biological systems, bridging it with molecular pharmacology. The present study is especially designed to explore biomarkers and tools for early diagnosis of diabetes mellitus type 2 with objective Western markers and TCM.

Objectives: The primary objective of the present study is to determine consistency in classification of DM type 2 in three categories as defined by Traditional Chinese Medicine (TCM) in pre-diabetic subjects.

Secondary objectives are to find relationships between diagnosis according to TCM and risk profile according to Western approach (fasting glucose and HbA1c in plasma, age, BMI, waist circumference). Another objective is to find relationships between classification of risk for DM type 2 according to TCM and objective parameters.

Study design: This study is designed as an explorative study. Study population: In the study 50 pre-diabetic male volunteers, with a fasting blood glucose ≥ 6.1 and ≤ 6.9 mmol/L, 30-70 years old, and having a BMI ≥ 26 and ≤ 35 kg/m2 will participate.

Intervention: No administration of a study substance will take place.

Main study parameters/endpoints:

TCM Diagnosis:Identification of DM type 2 based on TCM, diagnosed independently by 3 physicians and classified in Upper Xiao, Middle Xiao and Lower Xiao.

General measurements as BMI, waist circumference, blood pressure and heart rate variability will be conducted.

Next to these measurements also the following parameters will be established. Biophoton emission: a recording of the energy field and balance based on analysis of intensity and quantum stochastic nature of light from both hands (ventral and dorsum), in combination with both right-left and dorsal-ventral symmetry of both hands.

Performance Meridian Measurements (MERID measurements): The 'MERID' meridian method is based on the change of skin impedance after a given IR (infrared) stimulus to a Biological Active Point (BAP) which gives a reliable and reproducible measure for the energy status of that particular meridian and consequently of the related organ or organ system.

Heart rate variability:

Heart rate is affected by both sympathetic and parasympathetic input. These two branches of the autonomic control system affect both heart rate and changes in heart rate. Cardiac autonomic balance, also called sympatho-vagal balance, is the combined effect of parasympathetic (inhibitory) and sympathetic (excitatory) innervation of the heart and can be considered the main determinant of the regulation of heart rate and can be quantified by means of electrocardiography (ECG) measurements and spectral analysis.

Metabolomics:

Metabolomics to be applied in this study consists of a number of methods based on LC-MS and GC-MS technology to determine (relative) concentrations of endogenous metabolites in biological samples (blood and urine).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

This study is set up as a study with an explorative character. No administration of substances will take place. All subjects will be subjected to seven non-invasive measurements, filling in a number of questionnaires and subjected to three physical examinations. Blood sampling, in the fasting state, will be done at two determined time points (pre-study and in study) and will not exceed 30 mL. Furthermore, one (spot) urine sample will be collected in the study.

Based on the above mentioned assessments and the fact that no administration of substances will take place, the discomfort for the subjects in the study is minimal and the risk for participating subjects is negligible.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as assessed by the

   * health and lifestyle questionnaire, (P7348 F02; in Dutch)
   * physical examination
   * results of the pre-study laboratory tests
2. Males aged between 30 and 70 years at Day 01 of the study
3. Body Mass Index (BMI) between 26 and ≤ 35 kg/m2
4. Pre-diabetic as established by fasting glucose 6.1 to 6.9 mmol/L
5. Normal Dutch eating habits as assessed by P7348 F02
6. Voluntary participation
7. Having given written informed consent
8. Willing to comply with the study procedures
9. Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data for at least 15 years
10. Willing to accept the disclosure of the financial benefit of participation in the study to the authorities concerned

Exclusion Criteria:

1. Participation in any clinical trial including blood sampling and/or administration of substances up to 90 days before Day 01 of this study
2. Participation in any non-invasive clinical trial up to 30 days before Day 01 of this study, including no blood sampling and/or oral, intravenous, inhalatory administration of substances
3. Having a history of medical or surgical events that may significantly affect the study outcome
4. Medication use
5. Smoking
6. Alcohol consumption > 28 units/week
7. Reported unexplained weight loss or gain of > 2 kg in the month prior to the pre-study screening
8. Reported slimming or medically prescribed diet
9. Reported vegan, vegetarian or macrobiotic
10. Acupuncture treatment or use of TCM
11. Recent blood donation (<1 month prior to the start of the study)
12. Not willing to give up blood donation during the study
13. Personnel of TNO Quality of Life, their partner and their first and second degree relatives
14. Not having a general practitioner
15. Not willing to accept information-transfer concerning participation in the study, or information regarding his/her health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner.

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-06; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilrike J Pasman, PhD, Principal Investigator — TNO
Locations (1):
- Metabolic ward of TNO Quality of Life, Zeist, Utrecht, Netherlands